CLINICAL TRIAL: NCT00719615
Title: The Relationship Between Vitamin D and Thyroid Cancer
Brief Title: Assess Vitamin D Levels in Those With & Without Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0136-08-EP
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Thyroid Nodules; Vitamin D
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Thyroid Cancer in Remission Group: Thyroid Cancer-Remission Group & use of Vitamin D
- Thyroid Cancer with Active Disease Group: Thyroid Cancer-Active Group & use of Vitamin D
- Thyroid nodule group (no cancer) & Vit D: Thyroid nodule group without cancer and use of Vitamin D

SUMMARY:
The purpose of this study is to evaluate Vitamin D levels in thyroid cancer patients with active disease compared with thyroid cancer patients in remission and patients with thyroid nodules.

DETAILED DESCRIPTION:
Thyroid cancer is the most common endocrine related malignancy, increasing in incidence in recent years. There are relatively few, well known factors, both genetic and environmental, which predispose to the development of thyroid cancer. Vitamin D deficiency has been associated with other cancers, but the association between vitamin D and thyroid cancer is unknown. We plan to do a case control, pilot study to evaluate the relationship between vitamin D levels and thyroid nodules, thyroid cancer in remission, and active thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cases: History of Papillary, Follicular, Follicular Variant of Papillary, or Hurthle cell thyroid cancer (both active disease and in remission).
* Controls: Individuals with a thyroid nodule, matched to cases for age, BMI, season of vitamin D measurement.
* Participating in University of Nebraska Medical Center Thyroid Tumor and Cancer Collaborative Registry database.

Exclusion Criteria:

* Pregnant or breast feeding women
* Medullary thyroid cancer
* Anaplastic thyroid cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Thyroid Tumor and Cancer Collaborative Registry (TCCR) is a thyroid cancer and thyroid nodule database at the University of Nebraska Medical Center. The database serves as a registry and biospecimen bank for those who wish to participate in multidisciplinary research. The database will be accessed to query for individuals with a diagnosis of thyroid cancer, both active disease and in remission, as well as a diagnosis of thyroid nodules. Those meeting eligibility requirements will then have their registry information and stored biospecimens accessed for testing and review.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2008-05-28 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan W Laney, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] National Cancer Institute 2006 Handbook, National Cancer Institute, Bethesda, MD. http://obf.cancer.gov/financial/attachments/06Factbk.pdf.
- [Background] Garland CF, Garland FC, Gorham ED, Lipkin M, Newmark H, Mohr SB, Holick MF. The role of vitamin D in cancer prevention. Am J Public Health. 2006 Feb;96(2):252-61. doi: 10.2105/AJPH.2004.045260. Epub 2005 Dec 27. PMID 16380576
- [Background] Lappe JM, Travers-Gustafson D, Davies KM, Recker RR, Heaney RP. Vitamin D and calcium supplementation reduces cancer risk: results of a randomized trial. Am J Clin Nutr. 2007 Jun;85(6):1586-91. doi: 10.1093/ajcn/85.6.1586. PMID 17556697
- [Background] Ahonen MH, Tenkanen L, Teppo L, Hakama M, Tuohimaa P. Prostate cancer risk and prediagnostic serum 25-hydroxyvitamin D levels (Finland). Cancer Causes Control. 2000 Oct;11(9):847-52. doi: 10.1023/a:1008923802001. PMID 11075874
- [Background] Abbas S, Linseisen J, Slanger T, Kropp S, Mutschelknauss EJ, Flesch-Janys D, Chang-Claude J. Serum 25-hydroxyvitamin D and risk of post-menopausal breast cancer--results of a large case-control study. Carcinogenesis. 2008 Jan;29(1):93-9. doi: 10.1093/carcin/bgm240. Epub 2007 Oct 31. PMID 17974532
- [Background] Krishnan AV, Moreno J, Nonn L, Malloy P, Swami S, Peng L, Peehl DM, Feldman D. Novel pathways that contribute to the anti-proliferative and chemopreventive activities of calcitriol in prostate cancer. J Steroid Biochem Mol Biol. 2007 Mar;103(3-5):694-702. doi: 10.1016/j.jsbmb.2006.12.051. Epub 2007 Jan 16. PMID 17229571
- [Background] Welsh J. Vitamin D and prevention of breast cancer. Acta Pharmacol Sin. 2007 Sep;28(9):1373-82. doi: 10.1111/j.1745-7254.2007.00700.x. PMID 17723171
- [Background] Liu W, Asa SL, Fantus IG, Walfish PG, Ezzat S. Vitamin D arrests thyroid carcinoma cell growth and induces p27 dephosphorylation and accumulation through PTEN/akt-dependent and -independent pathways. Am J Pathol. 2002 Feb;160(2):511-9. doi: 10.1016/S0002-9440(10)64870-5. PMID 11839571
- [Background] Dackiw AP, Ezzat S, Huang P, Liu W, Asa SL. Vitamin D3 administration induces nuclear p27 accumulation, restores differentiation, and reduces tumor burden in a mouse model of metastatic follicular thyroid cancer. Endocrinology. 2004 Dec;145(12):5840-6. doi: 10.1210/en.2004-0785. Epub 2004 Aug 19. PMID 15319350
- [Background] Khadzkou K, Buchwald P, Westin G, Dralle H, Akerstrom G, Hellman P. 25-hydroxyvitamin D3 1alpha-hydroxylase and vitamin D receptor expression in papillary thyroid carcinoma. J Histochem Cytochem. 2006 Mar;54(3):355-61. doi: 10.1369/jhc.5A6734.2005. Epub 2005 Nov 28. PMID 16314444
- See also: SEER Database. — http://seer.cancer.gov/.
- See also: National Cancer Institute 2006 Handbook, National Cancer Institute, Bethesda, MD. http:// — http://obf.cancer.gov/financial/attachments/06Factbk.pdf.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals (at University of Nebraska Medical Center)were selected from a thyroid tumor and cancer collaborative registry (TCCR), database & biospecimen bank, started March 2008. We achieved a sample size of 111 subjects with 24 patients with active thyroid cancer, 45 patients with thyroid cancer in remission and 42 patients with thyroid nodules.
Pre-assignment Details: Individuals who had agreed to participate in the TCCR and who had also given a blood sample were included in sequential order.
Period: Overall Study
Arm/Group | Thyroid Nodules | Thyroid Cancer in Remission | Active Thyroid Cancer
Started | 42 | 45 | 24
Completed | 42 | 45 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thyroid Nodules | Thyroid Cancer in Remission | Active Thyroid Cancer | Total
Number analyzed (Participants) | 42 | 45 | 24 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 44 | 22 | 106
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 17 | 94
  Male | 4 | 6 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 42 | 45 | 24 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Persons That Are Vitamin D Deficient in the Thyroid Nodule, Thyroid Cancer in Remission, and the Active Thyroid Cancer Groups.
Description: We evaluated serum calcium,creatinine,albumin,and 25-hydroxyvitaminD(25-OH-D)in 42 thyroid nodule, 45 thyroid cancer in remission, & 24 active thyroid cancer patients. We also determined the number and percent of participants in each group that had vitamin D deficiency, defined as 25-OH-D < 30 ng/ml.
Time Frame: Within 12 months of enrollment in thyroid cancer collaborative registry (TCCR) database
Population: This study is a pilot study to provide preliminary data. Per protocol, we accrued 37% of the sample size needed for a fully powered study. Using the outcome "the proportion of persons with "vitamin D deficiency", a sample size of 160 subjects (64 nodule, 64 remission, and 32 active) would achieve an 80% power to detect an effect size of 0.25.
Measure: Number; unit: participants
Arm/Group | Thyroid Nodules | Thyroid Cancer in Remission | Active Thyroid Cancer
Number analyzed (Participants) | 42 | 45 | 24
participants | 23 | 20 | 11
Statistical Analysis 1: Comparison: Thyroid Nodules; Patient characteristics for each group were assessed using descriptive statistics, including medians, range, frequencies, and proportions. Categorical outcomes were compared between the 3 groups using a Fisher's exact test. A logistic regression modeling procedure was used to compare the odds of a low vitamin D levels between patient groups while adjusting for other risk factors: gender, age, BMI, season, and TNM staging; Test type: Superiority or Other; p < 0.05, Fisher Exact — Only risk factors significant at the 0.10 level in univariate analysis were included in the multivariate model

ADVERSE EVENTS:
Time Frame: breach of confidentiality
Description: This is a study evaluating stored blood from an established biobank. There was no risk to the patient, except the potential breach of confidentiality.
Arm/Group | Thyroid Nodules | Thyroid Cancer in Remission | Active Thyroid Cancer
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45 | 0/24
Other Adverse Events (participants affected / at risk) | 0/42 | 0/45 | 0/24

LIMITATIONS AND CAVEATS:
The trial limitations include that it was mostly done on Caucasian subjects; the controls were those with thyroid nodules not subjects without any thyroid disease; the sample size was small; & a small number of Vit D assays used different methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No